CLINICAL TRIAL: NCT04695041
Title: A Phase 1, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of PBI-4050 in Healthy Subjects
Brief Title: A Healthy Volunteer Study of PBI-4050
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Liminal BioSciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PBI-4050-CT-9-20
Record Dates: First submitted 2020-12-16; First posted 2021-01-05 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Fibrosis; Inflammation
MeSH Terms: conditions — Fibrosis; Inflammation | interventions — setogepram

STUDY DESIGN:
Intervention Model Description: Cohorts will be dosed sequentially in an ascending fashion with approximately 14 days between starting dose at each dose level.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort A: 1200 mg PBI-4050 (Experimental)
  Interventions: Drug: PBI-4050/ Placebo
- Cohort B: 1600 mg PBI-4050 (Experimental)
  Interventions: Drug: PBI-4050/ Placebo
- Cohort C: 2000 mg PBI-4050 (Experimental)
  Interventions: Drug: PBI-4050/ Placebo
- Cohort D: 2400 mg PBI-4050 (Experimental)
  Interventions: Drug: PBI-4050/ Placebo
- Cohort E: 2400 mg PBI-4050 (Experimental)
  Interventions: Drug: PBI-4050/ Placebo
- Cohort F (Supplemental): 1600 mg PBI-4050 (Experimental)
  Interventions: Drug: PBI-4050/ Placebo

INTERVENTIONS:
Drug: PBI-4050/ Placebo — Participants receive either 800mg PBI-4050 capsules or placebo, twice a day for 14 days
  Arms: Cohort B: 1600 mg PBI-4050; Cohort F (Supplemental): 1600 mg PBI-4050
Drug: PBI-4050/ Placebo — Participants receive either 1200mg PBI-4050 capsules or placebo, once a day for 14 days
  Arms: Cohort A: 1200 mg PBI-4050
Drug: PBI-4050/ Placebo — Participants receive either 1000 mg PBI-4050 capsules or placebo, twice a day for 14 days
  Arms: Cohort C: 2000 mg PBI-4050
Drug: PBI-4050/ Placebo — Participants receive either 1200 mg PBI-4050 capsules or placebo, twice a day for 14 days
  Arms: Cohort D: 2400 mg PBI-4050
Drug: PBI-4050/ Placebo — Participants receive either 800 mg PBI-4050 capsules or placebo, three times a day for 14 days
  Arms: Cohort E: 2400 mg PBI-4050

SUMMARY:
The purpose of this study is to investigate the study drug PBI-4050 to determine the safety, tolerability and concentration profile in the blood when the drug is given to healthy volunteers as multiple doses and different dosing regimens over a period of 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female of non-childbearing potential, between ≥18 years and ≤65 years of age, inclusive, at screening.
2. Female subject of non-childbearing potential. For the purposes of this study, this is defined as the subject being amenorrhoeic for at least 12 consecutive months prior to study drug administration or at least 6 months post-surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy).
3. Female subject with a negative pregnancy test at screening and admission.
4. Male subject (and partner of childbearing potential) willing to use a highly effective method of contraception or 2 effective methods of contraception, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of the investigation medicinal product (IMP).
5. Male subjects (including men who have had vasectomies) with a pregnant partner must agree to use a condom from first dose until at least 3 months (90 days) after last dose of IMP.
6. Male subjects must be willing to not donate sperm until 3 months (90 days) following last dose of IMP.
7. Subject with a body mass index (BMI) of >18.5 and <30 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females (BMI = body weight (kg) / [height (m)]2), at screening.
8. Healthy as defined by:

   1. Absence of clinically significant illness and surgery within 4 weeks prior to dosing. Subjects vomiting within 24 hours (h) pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the PI.
   2. Absence of clinically significant history of neurological, endocrinal, cardiovascular, pulmonary, haematological, immunologic, psychiatric, gastrointestinal, renal, hepatic and metabolic disease.
9. Continuous non-smoker who has not used tobacco or nicotine-containing products for at least 3 months prior to Screening and throughout the study, or users of cigarette replacements (i.e., e-cigarettes, nicotine patches or gums).
10. No clinically significant history of previous allergy / sensitivity to PBI-4050 or any of the excipients contained within the IMP(s).
11. No clinically significant abnormal test results for serum biochemistry, haematology, coagulation, and/or urine analyses within 28 days before the first dose administration of the IMP.
12. Subject with a negative urinary drugs of abuse (DOA) screen (including cotinine) and alcohol breath test results, determined within 28 days before the first dose administration of the IMP (N.B.: A positive alcohol and/or cotinine test result may be repeated at the Investigator's discretion).
13. Subject with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) and hepatitis C virus antibody (HCV Ab) test results at screening.
14. Subject must be available to complete the study (including all follow up visits).
15. Subject must satisfy an Investigator about his/her fitness to participate in the study.
16. Subject must provide written informed consent to participate in the study.

Exclusion Criteria:

1. A clinically significant abnormality or abnormal laboratory test results found during medical screening or a positive test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) found during medical screening.
2. Evidence of clinically significant hepatic or renal impairment including alanine aminotransferase (ALT) and aspartate aminotransferase (AST) above 1.2 x the upper limit of normal (ULN), direct bilirubin above 1.2 x ULN (total bilirubin accepted up to 2 x ULN if direct bilirubin is within normal limits), or creatinine is above ULN.
3. An estimated creatinine clearance as assessed by the Cockroft-Gault equation <60 mL/min at screening or admission.
4. Positive urine drug screen (including cotinine) or alcohol breath test at Screening or admission.
5. History of significant allergic reactions (e.g. anaphylactic reaction and angioedema) to any drug.
6. Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to the first study drug administration.
7. Female subject with a positive pregnancy test at screening or admission.
8. Clinically significant electrocardiogram (ECG) abnormalities at screening or admission, including PR > 220ms QTcF > 450ms.
9. Supine / Semi-supine systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg at screening.
10. Heart rate less than 40 or over 100 bpm at screening or admission.
11. A clinically significant history of drug or alcohol abuse [defined as the consumption of more than 14 units for male and female subjects) of alcohol a week], including use of soft drugs (such as marijuana) or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin and amphetamine derivatives) within the past year.
12. Participation in a New Chemical Entity (NCE) clinical study within the previous 3 months or a marketed drug clinical study within the 30 days before the first dose of IMP, or administration of a biological product in the context of a clinical research study within the 90 days before the first dose of IMP or concomitant participation in an investigational study involving no drug or device administration. (Washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
13. Use of medication other than topical products without significant systemic absorption, unless in the opinion of the Investigator and Sponsor's Responsible Physician the medication will not interfere with the study procedures or compromise subject safety:

    1. Prescription medication within 14 days prior to dosing;
    2. Non-prescription medication including vitamins, herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer), and ibuprofen within 48 h prior to the first dose of IMP,
    3. A depot injection or an implant of any drug within 3 months before the first dose of IMP.
14. Donation of 450 mL or more blood within the 3 months before the first dose of IMP.
15. Donation of plasma within 7 days prior to dosing.
16. Receipt of blood products within 2 months prior to admission.
17. Haemoglobin <130 g/L (males) and <115 g/L (females) and haematocrit <0.36 L/L (males) and <0.32 L/L (females) at screening or admission.
18. Breast feeding or lactating female subject.
19. A clinically significant history of gastrointestinal disorder likely to influence IMP absorption.
20. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
21. Inability to communicate well with the Investigators (i.e., language problem, poor mental development or impaired cerebral function).
22. Subjects with any special food restrictions that would hinder ability to consume the high fat breakfast provided during the study; e.g. vegetarian, lactose intolerance, vegan, low-fat, low sodium, and/or restrictions for medical, religious, social or cultural reasons, etc).
23. Any reason which, in the opinion of the PI, would prevent the subject from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Day 1 - Day 23 +/- 2 days
  Number and Severity of Treatment Emergent Adverse Events

SECONDARY OUTCOMES:
AUC | Day 1 and Day 14
  Area under PK curve
Cmax | Day 1
  Maximum plasma concentration (Cmax)
Cmax ss | Day 14
  Maximum steady-state plasma drug concentration during a dosage interval (Cmax ss)

CONTACTS AND LOCATIONS:
Locations (1):
- Covance CRU, Ltd., Leeds, United Kingdom